CLINICAL TRIAL: NCT00770367
Title: Pioglitazone and Serum Asymmetric Dimethylarginine (ADMA) in Patients With Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Takeda 07-060; 18379 (Other: IRB)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2011-12

CONDITIONS: Diabetes
Keywords: Cardiovascular risk; biological markers
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone then Placebo (Experimental): 18 volunteers that are Diabetic adults, 40-75 years that have higher ADMA levels as well as increased inflammation will take Pioglitazone for the first 12 week period of the study and then take the placebo for the final 12 weeks of the study.
  Interventions: Drug: Pioglitazone then Placebo
- Placebo then Pioglitazone (Experimental): 18 (other half of participants) volunteers that are Diabetic adults, 40-75 years that have higher ADMA levels as well as increased inflammation will take the placebo for the first 12 week period of the study and then take the Pioglitazone for the final 12 weeks of the study.
  Interventions: Drug: Placebo then Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone then Placebo — Subjects will take the pioglitazone 30mg tablet daily for 3 months. This will be followed by a 4-week period during which subjects will not be taking either the study drug or placebo. During the final 12-week period the group will take a placebo.
  Other Names: Actos, Glustin, Zactos
  Arms: Pioglitazone then Placebo
Drug: Placebo then Pioglitazone — Subjects will take the placebo for the first 12 weeks of the study. This will be followed by a 4-week period during which subjects will not be taking either the study drug or placebo. During the final 12-week period the group will take the pioglitazone 30mg tablet daily for 3 months.
  Other Names: Actos, Glustin, Zactos
  Arms: Placebo then Pioglitazone

SUMMARY:
SPECIFIC AIMS

1. To determine whether pioglitazone will reduce levels of asymmetric dimethylarginine(ADMA) in patients with diabetes.
2. To determine whether nitric oxide(NOx) products are increased with pioglitazone treatment.
3. To determine whether pioglitazone reduces oxidative stress (F2-isoprostanes).

DETAILED DESCRIPTION:
The primary purpose of this study is to determine whether treatment with pioglitazone can reduce serum levels of asymmetric dimethylarginine (ADMA) in patients with adult diabetes. Recent research has found that elevated serum ADMA is associated with increased cardiovascular events and mortality, particularly in people with diabetes (Boger 2005, Zoccali 2006, Ueda 2007). ADMA, by mediating nitric oxide (NO) availability, may trigger pro-atherogenic effects. High plasma concentration of this substance has been associated with intima-media thickening, left ventricular hypertrophy and all-cause and cardiovascular mortality in patients with end-stage renal disease, and associated with increased cardiovascular events in patients with diabetes (Kryzazanowska 2007). The result of higher levels of ADMA and reduced output of NO increases vasoconstriction, increases inflammation, and interferes with endothelial function. Preliminary studies indicate that pioglitazone may reduce ADMA levels, and thus lower cardiovascular risk.Thus, this protocol will test whether pioglitazone can reduce ADMA levels in adult patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 40--75 years-of-age, non-pregnant
* Informed consent
* History of type 2 Diabetes Mellitus
* Stable weight for the last 3 months (no change greater than +5% of body weight)
* ADMA > 0.50 µM/L (mean of non-diabetic reference group) (Devangelio 2007)
* On stable medical therapy for at least 3 months
* A working telephone

Exclusion Criteria:

* Any history of known coronary heart disease, including a history of congestive heart failure, myocardial infarction, coronary re-vascularization, or stroke
* Pregnancy
* Chronic kidney disease, serum creatinine >2.0mg/dl, chronic liver disease, or uncontrolled hypertension (>160/100).
* Current participation in a formal weight loss program or planning to start such a program during the next 3 months
* Collagen vascular disease, infection, or other inflammatory condition
* Electrocardiogram (EKG) evidence of ischemia or infarction
* Macular edema (swelling of the back of the eye), recent excessive weight gain (over 5% of weight in 30 days), elevated liver function tests > 2.5 X the upper limit, or history of osteoporosis

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana E King, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Department of Family Medicine, MUSC, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic, 36 participants recruited
Pre-assignment Details: After informed consent, a laboratory specimen will be obtained at the visit, including a pregnancy test (if indicated), and the screening ADMA level. This information will be used to determine study eligibility. Screened participants will be eligible if their ADMA > 0.50 μM/L. If not eligible would be excluded from study.
Groups:
- Pioglitazone: This is the analysis period during which participants took Pioglitazone.
- Placebo: The analysis period during which participant took the placebo.
Period: First Intervention
Arm/Group | Pioglitazone | Placebo
Started | 18 | 18
Completed | 18 | 16
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Washout Period of 4 Weeks
Arm/Group | Pioglitazone | Placebo
Started | 18 | 16
Completed | 18 | 15
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Pioglitazone | Placebo
Started | 18 | 15
Completed | 16 | 15
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (1.89) | 55.7 (2.42) | 54 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Asymmetric Dimethylarginine (ADMA) Level
Description: Labs measured micro moles per liter of ADMA levels in participants.
Time Frame: 3 months
Population: Recruited 36 participants per randomization.1st analysis is serum Asymmetric Dimethylarginine ADMA at 12 weeks b/w groups.
Measure: Mean (95% Confidence Interval); unit: umol/L
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 36 | 36
umol/L | .80 [.75 to .85] | .75 [.71 to .79]
Statistical Analysis 1: Comparison: Pioglitazone vs Placebo; A twosample comparison of mean treatment differences conducted using a pre-determined significance level of alpha level <0.05. 2 a comparison of means for NOx levels at 12 weeks b/w groups. 3 on the change F2-isoprostanes at 12 weeks b/w groups; Test type: Non-Inferiority or Equivalence — Equivalence; p = .37, t-test, 2 sided; Mean Difference (Final Values) = .05, Standard Error of Mean .05

2. Secondary Outcome: NOx f2-isoprostanes
Description: Measured oxidative stress - NOx measured by chemiluminescence detection using the Sievers NOA 280i and f2-isoprostanes are isolated by thin layer chromatography and subjected to a highly sensitive and specific gas chromatography/mass spectroscopy method to measusre the oxidative stress
Time Frame: 3 months
Population: 36 adults with diabetes enrolled in the study, and 31 completed the 7-month protocol. Adherence with medication was 93% during the trial according to pill counts at the final visit. Participants were allowed to take their other regular medications during the trial.
Measure: Mean (Standard Error); unit: Oxidative stress
Arm/Group | Pioglitazone Then Placebo | Placebo Then Pioglitazone
Number analyzed (Participants) | 18 | 18
Oxidative stress | -1.4 (1.4) | -1 (2.6)

ADVERSE EVENTS:
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No